CLINICAL TRIAL: NCT06569316
Title: Journey to Understanding - Indigenous Peoples Engagement in Cancer Research Arizona (JUNIPER)
Brief Title: Genetic Testing for the Prevention of Cancer in Indigenous American Communities (JUNIPER Trial)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 24-006285; NCI-2024-06870 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-006285 (Other: Mayo Clinic Institutional Review Board); MC240902 (Other: Mayo Clinic in Arizona); U2CCA252973 (NIH)
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Specimen Handling; Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (blood, saliva, tissue collection, genetic testing) (Experimental): Patients undergo collection of blood or saliva samples on study for genetic testing. Patients also undergo collection of leftover tissue obtained from SOC surgical procedure or biopsy, or stored tissue samples for genetic testing on study. Patients receive the results of their genetic testing and are given resources for counseling and further care.
  Interventions: Procedure: Biospecimen Collection; Other: Communication Intervention; Other: Genetic Testing; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood or saliva and leftover tissue sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Communication Intervention — Receive care plan recommendations
Other: Genetic Testing — Undergo genetic testing
  Other Names: Genetic Analysis; Genetic Examination; Genetic Test
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial is studying the genetic changes in cells associated with different types of cancer in Indigenous American (IA) populations in the Southwest to improve cancer screening, precision prevention, and therapeutic intervention for individual in these communities. IA tribes have much lower rates of cancer screening, have more limited access to healthcare, are more often diagnosed at later stages of disease, and have the poorest outcomes in all types of cancer when compared to any other racial and ethnic group in the United States. Due to these significant cancer health disparities, IAs have been understudied and little is known about the molecular characterization of tumors arising in IAs. Undergoing genetic testing of tumors may improve cancer outcomes in IA participants and communities.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop culturally appropriate, respectful, trusted, and collaborative means to engage and recruit Indigenous Americans (IAs) affected by cancer (newly diagnosed cancer participants, participants undergoing cancer treatment, and cancer survivors) for molecular characterization of their tumors.

Ia. Conduct direct participant engagement with cancer participants/survivors, community advisors, and partners to refine and optimize methods/processes.

Ib. Identify, recruit, and consent eligible IA cancer participants/survivors. Ic. Implement tissue acquisition, epidemiologic, behavioral, and clinical data collection, conduct continuous assessment of performance benchmarks.

Id. Return clinical grade and clinically useful genomic data to participants with navigation to counseling and clinical resources as warranted and as they select.

SECONDARY OBJECTIVE:

I. Translate any discoveries to improved cancer screening, precision prevention, and therapeutic intervention that can be used to enhance cancer screening and precision prevention and improve cancer outcomes in Indigenous American participants and communities.

OUTLINE:

Patients undergo collection of blood or saliva samples on study for genetic testing. Patients also undergo collection of leftover tissue obtained from standard of care (SOC) surgical procedure or biopsy, or stored tissue samples for genetic testing on study. Patients receive the results of their genetic testing and are given resources for counseling and further care.

After completion of study intervention, patients are followed up once a year up to 5 years from study registration.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults >= 18 years of age
* Cancer patient undergoing active treatment or a cancer survivor
* Self-identify as Indigenous American

Exclusion Criteria:

* Unable to provide informed consent
* Individuals who are under 18 years of age
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Successful accrual of Indigenous American (IA) participants | Up to 5 years
  Assessed by the number of IA participants consented to study.
Return of valuable genetic results to participants | Up to 5 years
  Assessed by the number of participants who receive genetic results. Clinically useful genomic data will be returned to participants with navigation to counseling and clinical resources as warranted and as they select.

CONTACTS AND LOCATIONS:
Overall Officials: Jewel Samadder, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials